CLINICAL TRIAL: NCT00936871
Title: A Phase 1, Randomized, Single Dose, Placebo And Active Controlled, 3-Way Crossover Study To Evaluate The Effect Of A Single Oral Dose Of Lersivirine (UK-453,061) On Qt Intervals In Healthy Subjects
Brief Title: The Effect Of Lersivirine (UK-453,061) On Qt Intervals In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A5271032
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
Keywords: lersivirine QT QTc ECG HIV NNRTI
MeSH Terms: interventions — UK 453,061; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Lersivirine Tolerability
  Interventions: Drug: Lersivirine; Drug: Placebo; Drug: Lersivirine (if necessary)
- Part B (Experimental): Thorough QTc
  Interventions: Drug: Lersivirine; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Lersivirine — Lersivirine 2400 mg single dose
  Arms: Part A
Drug: Placebo — Placebo single dose
  Arms: Part A
Drug: Lersivirine (if necessary) — Lersivirine 2100 mg single dose (if necessary)
  Arms: Part A
Drug: Lersivirine — Lersivirine 2400 mg single dose (dose may be decreased pending Part A tolerability results)
  Arms: Part B
Drug: Placebo — Placebo single dose
  Arms: Part B
Drug: Moxifloxacin — Moxifloxacin 400 mg single dose
  Arms: Part B

SUMMARY:
This study has been designed to investigate the effect of lersivirine on the QT/QTc interval in order to help establish the safety profile of lersivirine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive, (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, normal 12-lead ECG and clinical laboratory tests)

Exclusion Criteria:

* History of risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesemia, congenital long QT syndrome, myocardial ischemia or infarction).
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
(Part A) To evaluate the safety and toleration of a single dose of lersivirine in healthy male and female subjects. | 1 day
(Part B) To demonstrate a lack of effect of lersivirine on QTc relative to time-matched placebo. | 3 days

SECONDARY OUTCOMES:
To determine study sensitivity by comparing the effect of moxifloxacin on QTc relative to time-matched placebo, at the historical moxifloxacin Tmax of 3 hours. | 1 day
To evaluate the safety and toleration of a single dose of lersivirine in healthy male and female subjects. | 1 day
To characterize the exposure-response relationship between lersivirine and changes in QTc using plasma concentrations of lersivirine. | 1 day
To assess the single dose pharmacokinetics of lersivirine. | 1 - 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271032&StudyName=The%20Effect%20Of%20Lersivirine%20%28UK-453%2C061%29%20On%20Qt%20Intervals%20In%20Healthy%20Subjects